CLINICAL TRIAL: NCT02924974
Title: Spinal Morphine in Robotic Assisted Radical Prostatectomy
Acronym: SALMON-RARP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L2015108
Record Dates: First submitted 2016-09-29; First posted 2016-10-05 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-03

CONDITIONS: Morphine; Injections, Spinal; Prostatectomy; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Morphine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): subcutaneous lidocaïne and intravenous loading dose of morphine
  Interventions: Drug: Lidocaine
- Intervention (Experimental): Spinal injection of 4 or 5 ml of bupivacaine/morphine 2,5 mg/ml/60mcg/ml. The reduction to 4 ml is for patients over 75 years of age
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — mixed with bupivacaine
  Arms: Intervention
Drug: Lidocaine — sham procedure (s.c. lidocaïne)
  Arms: Control

SUMMARY:
This study will investigate if a single shot of spinal morphine will increase patient satisfaction when compared to intravenous morphine in Robot-Assisted Radical Prostatectomy

DETAILED DESCRIPTION:
This study is a randomized controlled trial. It will randomize 160 patients who are scheduled for Robot-Assisted Radical Prostatectomy. The intervention group will receive a single spinal injection of a bupivacaine (12,5 mg)/morphine(300 mcg) mixture. Controlgroup will receive a subcutaneous injection of lidocaïne for placebo purposes and an intravenous loading dose of morphine at the end of surgery.

Both groups will receive general anesthesia during surgery in a standardized fashion.

After the surgery, both groups will receive a Patient-Controlled Analgesia pump for post-operative pain control.

Primary outcome is patient satisfaction as measured by the Quality-of-Recovery-15 questionnaire. This questionnaire will be taken at baseline, day 2 and 1 week after surgery.

Secundary outcomes are morphine use per PCA, duration of hospital stay, side-effects and ease of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Robot-Assisted Radical Prostatectomy

Exclusion Criteria:

* Contra-indications to spinal anesthesia (severe aortic stenosis, coagulation disorders)
* Contra-indications to study medication (local anesthetics, morphine, paracetamol, metamizol)
* Conversion to an open procedure
* Post-operative ICU-admission

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-05-25 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | day 1
  Quality of Recovery-15 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Seppe Koopman, MD, PhD, Study Chair — Maasstad Ziekenhuis; Aart Jan W Teunissen, MD, Study Chair — Maasstad Ziekenhuis; Mark V Koning, MD, DESA, Principal Investigator — Maasstad Ziekenhuis
Locations (1):
- Maasstad Hospital, Rotterdam, Netherlands

REFERENCES:
- [Derived] Koning MV, de Vlieger R, Teunissen AJW, Gan M, Ruijgrok EJ, de Graaff JC, Koopman JSHA, Stolker RJ. The effect of intrathecal bupivacaine/morphine on quality of recovery in robot-assisted radical prostatectomy: a randomised controlled trial. Anaesthesia. 2020 May;75(5):599-608. doi: 10.1111/anae.14922. Epub 2019 Dec 17. PMID 31845316